CLINICAL TRIAL: NCT04542876
Title: Efficacy and Safety of Guduchi Ghan Vati in the Management of Asymptomatic COVID-19 Infection: An Open Label Feasibility Study
Brief Title: Efficacy and Safety of Guduchi Ghan Vati in the Management of Asymptomatic COVID-19 Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarogyam UK (Other)
Collaborators: Dr. Sarvepalli Radhakrishnan Rajasthan Ayurved University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AYU/DSSR/03
Record Dates: First submitted 2020-09-08; First posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Amrita Bindu; guduchi

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ayurveda (Experimental): Guduchi Ghana is a unique Ayuvedic classical preparation prepared from aqueous extracts of Tinospora cordifolia stem.
  Interventions: Drug: Guduchi Ghan Vati

INTERVENTIONS:
Drug: Guduchi Ghan Vati — Guduchi Ghan Vati was orally administered 2 tablets (1000 mg) twice daily for 2 weeks.
  Other Names: Giloya; Amrita; Tinosporia Cordifolus; Guduchi

SUMMARY:
The emergence of asymptomatic patients poses a significant challenge to the prevention and treatment of the epidemic.There have not been any treatment options that reduce the viral load or preventive options that reduce the risk of developing severe conditions.Therefore, present feasibility study of the safety and efficacy of Guduchi Ghan Vati was conducted in asymptomatic patients with COVID-19

ELIGIBILITY:
Inclusion Criteria:

* All hospitalised cases above 18 years of age,
* Diagnosed with Covid-19
* Asymptomatic at the time of admission
* Agree to give consent

Exclusion Criteria:

* Symptoms relating to Covid-19
* Severe vomiting
* Respiratory failure or requiring mechanical ventilation
* Patients having alanine transaminase (ALT) or aspartate transaminase (AST) > 5 times the upper range of normal limits
* Patients with Covid-19 in critical condition or ARDS or NIAD 8 -point ordinal score-2
* Patients with uncontrolled diabetes mellitus
* Malignant,
* Chronic renal failure or
* On immunosuppressive medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-08-18 (Actual)

PRIMARY OUTCOMES:
Virologic clearance | 14 days
  Virologic clearance indicates the duration from the first Covid-19 positive result to the first Covid-19 negative result

SECONDARY OUTCOMES:
Hospital Stay | 14 days
  Total duration of stay in hospital for complete recovery
Clinically relevant adverse effects | 14 days
  Clinically relevant adverse effects of Guduchi Ghan Vati were reported using Adverse Drug Reaction reporting form
Laboratory tests | change from baseline to 14 days
  Routine blood tests were performed to assess complete blood counts, blood biochemistry parameters {Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Urea, C-reactive protein (CRP), as well as Albumin} and immunoglobulines.

CONTACTS AND LOCATIONS:
Overall Officials: Abhimanyu Kumar, Principal Investigator — Dr. Sarvepalli Radhakrishnan Rajasthan Ayurved University; Neha Sharma, Study Director — Aarogyam UK
Locations (1):
- Dr. Sarvepalli Radhakrishnan Rajasthan Ayurved University, Jodhpur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Undecided